CLINICAL TRIAL: NCT06516952
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis
Brief Title: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis (STOP-PN1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB54707-305; 2024-511879-16-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo nodularis; PN; INCB054707; chronic pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Povorcitinib Dose 1 (Experimental): Povorcitinib at the protocol-defined dose.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose 2 (Experimental): Povorcitinib at the protocol-defined dose.
  Interventions: Drug: Povorcitinib
- Placebo (Placebo Comparator): Placebo at the protocol-defined dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Povorcitinib — Oral Tablet
  Other Names: INCB054707
  Arms: Povorcitinib Dose 1; Povorcitinib Dose 2
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate effect of povorcitinib on itch and skin lesions in participants with prurigo nodularis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 to 75 years of age.
* Clinical diagnosis of PN for at least 3 months prior to Screening visit.
* Pruritus, defined as an average Itch NRS score ≥ 7 during the 7 days prior to Day 1/Baseline.
* Total of ≥ 20 pruriginous lesions on ≥ 2 different body regions (both legs, and/or both arms, and/or trunk) at Screening and Day 1/Baseline.
* Documented history of treatment failure, demonstrated intolerance, or contraindication to a previous PN treatment.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Chronic pruritus due to a condition other than PN or neuropathic and psychogenic pruritus.
* Diagnosis of PN secondary to medications.
* Active AD lesions (signs and symptoms other than dry skin) within 3 months prior to Screening visit.
* Women who are pregnant (or are considering pregnancy) or breastfeeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction; venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, stroke, moderate to severe heart failure, cerebrovascular accident, myocardial infarction, or other significant cardiovascular diseases; Q-wave interval abnormalities; disseminated herpes zoster or dermatomal herpes zoster; disseminated herpes simplex; chronic/recurrent infections; malignancies.
* Evidence of infection with TB, HBV, HCV or HIV.
* History of failure to any topical or systemic JAK or TYK2 inhibitor as treatment of PN or any inflammatory disease.
* Laboratory values outside of the protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Itch NRS4 and IGA-CPG-S-TS at Week 24 | Week 24
  Defined as proportion of participants achieving a ≥ 4-point improvement [reduction] in Itch NRS score from baseline (Itch NRS4) and an IGA CPG-S score of 0 or 1 with a ≥ 2-grade improvement from baseline (IGA-CPG-S-TS).

SECONDARY OUTCOMES:
Proportion of participants achieving Itch NRS4 at Week 24 | Week 24
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score from baseline.
Proportion of participants achieving IGA-CPG-S-TS at Week 24 | Week 24
  Defined as percentage of participants that achieve IGA-CPG-S score of 0 or 1 with a ≥ 2 grade improvement from baseline.
Proportion of participants achieving Itch NRS4 at Week 4 | Week 4
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score from baseline.
Time to Itch NRS4 | Up to 52 weeks
  Defined as time taken for the participant to achieve a ≥4 improvement in Itch NRS score from baseline.
Change from baseline in Itch NRS score at each postbaseline visit | Up to 52 weeks
  Itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Percent change from baseline in NRS score at each postbaseline visit | Up to 52 weeks
  Itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".
Proportion of participants achieving Itch NRS4 at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve a ≥ 4-point improvement in Itch NRS score from baseline.
Proportion of participants achieving IGA-CPG-S-TS at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve an IGA-CPG-S score of 0 or 1 with a ≥ 2 grade improvement from baseline.
Proportion of participants achieving Investigator's Global Assessment - Chronic Prurigo Activity (IGA-CPG-A) at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve an IGA-CPG-A score of 0 or 1 with a ≥ 2 grade improvement (reduction) from baseline.
Proportion of participants achieving ≥ 75% healed lesions in Prurigo Activity Score (PAS) at each postbaseline visit | Up to 52 weeks
  The modified PAS will be used in this study as defined by the protocol.
Proportion of participants achieving Itch NRS4 and IGA-CPG-S-TS at each postbaseline visit | Up to 52 weeks
  Defined as percentage of participants that achieve a ≥ 4-point improvement (reduction) in Itch NRS score and IGA-CPG-S score of 0 or 1 with a ≥ 2-grade improvement from baseline.
Change from baseline in Dermatology Life Quality Index (DLQI) score at each postbaseline visit. | Up to 52 weeks
  The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days.
Percent change from baseline in Dermatology Life Quality Index (DLQI) score at each postbaseline visit. | Up to 52 weeks
  The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days.
Proportion of participants with at least a 4-point decrease in DLQI score from baseline at each postbaseline visit for participants with DLQI score ≥ 4 at baseline | Up to 52 weeks
  Defined as percentage of participants with at least a 4-point decrease in DLQI score from baseline at each postbaseline visit for participants with DLQI score ≥ 4 at baseline.
Change from baseline in Skin Pain NRS score at each postbaseline visit | Up to 52 weeks
  Skin Pain NRS is an 11-point scale (0 to10) where 0 is "no pain" and 10 is the "worst pain imaginable".
Percent change from baseline in Skin Pain NRS score at each postbaseline visit | Up to 52 weeks
  Skin Pain NRS is an 11-point scale (0 to10) where 0 is "no pain" and 10 is the "worst pain imaginable".
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) score at each postbasline visit | Up to 52 weeks
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).
Percent change from baseline in the HADS score at each postbaseline visit | Up to 52 weeks
  HADS is a 14-item questionnaire that assesses the levels of anxiety and depression that a participant is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3).
Change from baseline in EQ-5D-5L score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Percent change from baseline in EQ-5D-5L score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score at each postbaseline visit | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Percent change in FACIT-F score at each postbaseline visit | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Proportion of participants with at least a ≥ 4-point increase in FACIT-F score at each postbaseline visit for participants with FACIT-F score ≤ 48 at baseline | Up to 52 weeks
  The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days.
Number of Participants with Treatment Emergent Adverse Events (TEAE) | Up to 52 weeks
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (120):
- United States (31):
  - Cahaba Dermatology, Birmingham, Alabama
  - Banner - University Medicine Multispecialty Services Clinic, Tucson, Arizona
  - Premier Dermatology Clinical Trials Institute At Northwest Arkansas, Fayetteville, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Northridge, Northridge, California
  - Rendon Center the Dermatology and Aesthetic Center, Boca Raton, Florida
  - Driven Research Llc, Coral Gables, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Research Institute of the Southeast, Llc, West Palm Beach, Florida
  - Illinois Dermatology Institute the Chicago Loop, Chicago, Illinois
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois
  - Center For Medical Dermatology and Immunology Research, Chicago, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Dermatology Specialists Research Ds Research Indiana Location, Clarksville, Indiana
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - The University of New Mexico Unm Health Sciences Center Hsc, Albuquerque, New Mexico
  - Montefiore Medical Center, East Syracuse, New York
  - Skin Center Dermatology Group, New York, New York
  - Stony Brook Dermatology Associates, Stony Brook, New York
  - Centricity Research Columbus, Columbus, Ohio
  - Wright State Physicians Health Center, Dayton, Ohio
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Sweetwater Dermatology, Sugar Land, Texas
  - Center For Clinical Studies, Webster, Texas
  - Frontier Dermatology, Mill Creek, Washington
- Argentina (7):
  - Conexa Investigacion Clinica S.A., Buenos Aires
  - Cedic - Consultorios Medicos, Buenos Aires
  - Instituto de Neumonologia Y Dermatologia, Buenos Aires
  - Instituto de Investigaciones En Alergia Y Enfermedades Respiratorias (Inaer), Buenos Aires
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto Especialidades de La Salud Rosario - Clinica Del Torax, Rosario
  - Investigaciones Reumatologicas Tucuman S.R.L., San Miguel de Tucumán
- Austria (2):
  - Medical University Graz University Clinic For Dermatology and Venerology, Graz
  - Wiener Krankenanstaltenverbund (Kav) - Krankenhaus Hietzing Mit Neurologischem Zentrum Rosenhuegel, Vienna
- Bulgaria (7):
  - Medical Center Medconsult Pleven, Lovech
  - Medconsult Pleven, Pleven
  - Diagnostic-Consultative Centre Pulmed Eood, Plovdiv
  - Medical Center Prolet Eood, Rousse
  - Medical Center Unimed Eood, Sevlievo
  - Diagnostic-Consultative Center Ascendent Eood, Sofia
  - Diagnostic-Consultative Center Aleksandrovska Eood, Sofia
- Canada (15):
  - Dermatology Research Institute, Calgary, Alberta
  - Rao Dermatology, Edmonton, Alberta
  - Skin Physicians, Edmonton, Alberta
  - Alpha Research-Lucere Dermatology and Laser Clinic, Edmonton, Alberta
  - Park Dermatology, Sherwood Park, Alberta
  - Simcoderm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Skin Health, Cobourg, Ontario
  - Centricity Research London Victoria Multispecialty, London, Ontario
  - Dermeffects, London, Ontario
  - North York Research Inc., Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Centre de Recherche Dermatologique de Quebec, Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Sima Recherche, Verdun, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- France (8):
  - Hopital Prive D Antony, Antony
  - Hospital Morvan, Brest
  - Cabinet Medical- Chemin de Paradis, Martigues
  - Ghrmsa Hopital Emile Muller, Mulhouse
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hopital Hotel Dieu, Nantes
  - Chu Paris-Gh St-Louis Lariboisiere F.Widal Hopital Saint-Louis, Paris
  - Hopitaux Drome Nord - Site de Romans Sur Isere, Romans-sur-Isère
  - Hopital Larrey, Toulouse
- Germany (13):
  - Aachen University Hospital, Aachen
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Hautzentrum Friedrichshain Studien, Berlin
  - Charite Universitatsmedizin Berlin, Berlin
  - Klinikum Dortmund Ggmbh, Dortmund
  - Universitaetsklinik Und Poliklinik Fuer Dermatologie Und Venerologie, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitatsklinik Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Schleswig-Holstein (Uksh) - Campus Luebeck, Lübeck
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitaetsklinikum Giessen Und Marburg Gmbh, Marburg
  - Universitaets-Hautklinik Eberhard-Karls-Universitaet Tuebingen, Tübingen
- Italy (9):
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico San Marco, Catania
  - Clinical Research Centre - Cast, Chieti
  - Azienda Sanitaria Locale 1 (Asl 1) - Ospedale Regionale San Salvatore, L’Aquila
  - Uoc Dermatologia Ospedale Maggiore Policlinico, Fondazione Irccs Ca' Granda, Milan
  - Aou Universita Della Campania Luigi Vanvitelli, Azienda Ospedaliero Universitaria Federico Ii Di Nap, Napoli
  - Azienda Ospedaliera Di Perugia, Perugia
  - Azienda Ospedaliero Universitaria Pisana - Ospedale S. Chiara, Pisa
  - Catholic University of the Sacred Heart, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
- Netherlands (2):
  - Amsterdam Umc Research Bv, Amsterdam
  - Maxima Medisch Centrum, Veldhoven
- Poland (15):
  - Niepubliczny Zaklad Opieki Zdrowotnej Specjalistyczny Osrodek Dermatologiczny Dermal, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Gyncentrum Sp. Z O.O., Nzoz Holsamed- Oddzial Libero, Katowice
  - Pro Familia Altera Sp. Z O.O., Katowice
  - Centrum Badan Klinicznych, Jagiellonskie Centrum Innowacji Sp.Z.O.O., Krakow
  - Diamond Clinic Sp. Z O.O., Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Med-Laser, Lublin
  - Mazowieckie Centrum Badan Klinicznych, Pruszków
  - Laser Clinic, Szczecin
  - Nzoz Gyncentrum - Oddzial Warszawa, Warsaw
  - Clinical Research Group Sp. Z.O.O, Warsaw
  - Centrum Medyczne Evimed, Warsaw
  - Klinika Ambroziak Sp. Z O.O., Warsaw
  - Dermaceum Centrum Badan Klinicznych, Wroclaw
  - Emc Instytut Medyczny Spolka Akcyjna-Euromedicare Szpital Specjalistyczny Z Przychodnia, Wroclaw
- South Korea (8):
  - Korea University Ansan Hospital, Ansan-si
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Pusan National University Hospital (Pnuh), Busan
  - Pusan National University Yangsan Hospital, Busan
  - The Catholic University of Korea, Incheon St. Mary'S Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
- Switzerland (3):
  - Inselspital Bern, Bern
  - Dsc Clinic Buochs, Buochs
  - Universitatsspital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Prurigo Nodularis (STOP-PN1) — https://incyteclinicaltrials.com/studies/incb54707-305